CLINICAL TRIAL: NCT05359016
Title: Evaluating Innovative Technologies and Approaches to Addressing Cervical Cancer in Gaza and Maputo Cidade Provinces in Mozambique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Population Services International (Other); Eduardo Mondlane University (Other); William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-0651; NCI-2022-03767 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-25; First posted 2022-05-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV testing of women for cervical cancer screening (Experimental): Women enrolled in this study will receive HPV testing for cervical cancer screening. They will be offered self-sampling. And also they will be offered voluntary Family Planning services, as appropriate.
  Interventions: Behavioral: HPV testing of women for cervical cancer screening

INTERVENTIONS:
Behavioral: HPV testing of women for cervical cancer screening — Women enrolled in this study will receive HPV testing for cervical cancer screening. They will be offered self-sampling. And also they will be offered voluntary Family Planning services, as appropriate.

SUMMARY:
The goal of this operational research study is to develop, implement and test integrated CCS&PT and voluntary FP service delivery models to evaluate whether integrated service delivery can optimize uptake and health impact of both services. The study objectives and learning questions are listed below, along with key outcomes that will be measured.

DETAILED DESCRIPTION:
Objectives:

The study objectives are outlined below:

1. To quantify the health impact of CCS&PT on the uptake of voluntary FP services.
2. To quantify the health impact of voluntary FP on the uptake of CCS&PT services.
3. To determine which promotional strategies are most effective to increase uptake of CCS&PT services.
4. To identify cost to deliver high quality CCS&PT services integrated into existing voluntary FP programs.
5. To determine client and provider acceptability of integrated CCS&PT and voluntary FP services using new screen and treat technologies.

ELIGIBILITY:
Inclusion Criteria:

* Women 30 - 49 years or all women living with HIV
* Not currently pregnant
* Patients with a cervix (women who have undergone a total hysterectomy with removal of the cervix are not eligible)
* Living in Maputo or Gaza
* Willing and able to provide informed consent for services.

Exclusion Criteria:

* Not meeting the inclusion criteria
* Physical or mental impairment that inhibits participation in the study
* Pregnant women

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 14600 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Number of women who will undergo Cervical Cancer Screening by HPV testing | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org